CLINICAL TRIAL: NCT01196377
Title: Personalized Medicine, Biomarker-based Study of Optimal Albuterol Regimens for Acute Asthma Exacerbations: DBRCT Pilot Study
Brief Title: Optimal Albuterol Regimens for Acute Asthma Exacerbations: DBRCT Pilot Study
Acronym: OARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Donald H Arnold, Associate Professor of Pediatrics and Emergency Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100725; K23HL080005 (NIH)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Acute Asthma
Keywords: Asthma; Acute asthma; Pediatrics
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nebulized albuterol 10mg/hr continuous (Active Comparator): Active control arm, 10mg/hr continuous.
  Interventions: Drug: Albuterol
- 10mg/hr pulsed (Experimental): Experimental 10mg/hr pulsed albuterol regimen.
  Interventions: Drug: Albuterol
- 25mg/hr continuous (Experimental): Experimental 25mg/hr continuous albuterol.
  Interventions: Drug: Albuterol
- 25mg/hr pulsed (Experimental): Experimental 25mg/hr pulsed albuterol
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: Albuterol — Nebulized albuterol
  Other Names: proventil

SUMMARY:
Our overall objective is to model a pediatric Acute Asthma Clinical Decision Rule (ADR) for personalized medicine by identification of treatment-response phenotypes that are important determinants of outcome. The Specific Aim of this study is to determine the feasibility of this approach by enrolling a pilot cohort of 16 participants in this DBRCT of 4 different albuterol treatment regimens, 2 of which will use 10mg/hr and 2 of which will use 25mg/hr. Within these dosages there will be a pulsed-treatment regimen and a continuous regimen.

DETAILED DESCRIPTION:
The objective of this study is to determine the feasibility of this approach by enrolling a pilot cohort of 16 participants in this DBRCT of 4 different albuterol treatment regimens, 2 of which will use 10mg/hr and 2 of which will use 25mg/hr. Participants are randomized in randomly permuted blocks of four. Within these dosages there will be a pulsed-treatment regimen and a continuous regimen.

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed asthma
* Acute asthma exacerbation
* Treatment with systemic corticosteroids and nebulized albuterol
* Ages 5 to 17 years

Exclusion Criteria:

* Other acute or chronic lung disease

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald H Arnold, MD, MPH, Principal Investigator — Vanderbilt University School of Medicine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 16 patients ages 5 to 17 years for this double blind randomized trial.
Groups:
- 25mg/hr Pulsed: Experimental 25mg/hr pulsed
Period: Overall Study
Arm/Group | Nebulized Albuterol 10mg/hr Continuous | 10mg/hr Pulsed | 25mg/hr Continuous | 25mg/hr Pulsed
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulized Albuterol 10mg/hr Continuous | 10mg/hr Pulsed | 25mg/hr Continuous | 25mg/hr Pulsed | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (2) | 7.9 (2) | 7.6 (4) | 7.7 (2) | 7.7 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 2 | 2 | 2 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: %FEV1
Description: % predicted forced expiratory volume in 1-second as a measure of airway obstruction
Time Frame: 2 hours
Measure: Mean (Full Range); unit: %-predicted
Arm/Group | Nebulized Albuterol 10mg/hr Continuous | 10mg/hr Pulsed | 25mg/hr Continuous | 25mg/hr Pulsed
Number analyzed (Participants) | 4 | 4 | 4 | 4
%-predicted
  Baseline, pretreatment | 20 [17 to 25] | 34 [19 to 41] | 26 [16 to 36] | 31 [14 to 41]
  2-hours (post-treatment) | 41 [32 to 48] | 47 [17 to 77] | 67 [61 to 73] | 44 [34 to 55]

ADVERSE EVENTS:
Time Frame: 2 hours
Description: Report is to data safety and monitoring committee and IRB.
Arm/Group | Nebulized Albuterol 10mg/hr Continuous | 10mg/hr Pulsed | 25mg/hr Continuous | 25mg/hr Pulsed
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Limitations: small sample size and not powered to detect differences in outcomes (pilot feasibility study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No